CLINICAL TRIAL: NCT04306666
Title: Early Rehabilitation After Hand or Wrist Ambulatory Surgery : How to Preserve Locomotion at Home Without Rebound Pain? Study Walant " Wide Awake Local Anesthesia No Tourniquet " Versus Axillary Brachial Plexus Block.
Brief Title: Early Rehabilitation After Hand or Wrist Ambulatory Surgery : How to Preserve Locomotion at Home Without Rebound Pain?
Acronym: WalantBAX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0429
Record Dates: First submitted 2019-11-29; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hand Surgery; Wrist Surgery
Keywords: Regional anesthesia; Walant block
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Walant group: Walant group
  Interventions: Other: Regional anesthesia
- Axillary Brachial Plexus Block: Axillary Brachial Plexus Block
  Interventions: Other: Regional anesthesia

INTERVENTIONS:
Other: Regional anesthesia — Injection of local anesthetics by a regional anesthesia named Walant block (Wide Awak Local anesthesia No Tourniquet)or by axillary brachial plexus block.

SUMMARY:
The purpose of this retrospective study is to compare the analgesic efficacy of Walant " Wide Awake Local Anesthesia No Tourniquet " with lidocaine and bupivacaine versus axillary brachial plexus block using mepivacaïne, both performed by anesthesiologists, after hand or wrist ambulatory surgery.

The main objective is to prove that Walant block improve pain relief at home measuring time to first analgesic request.

The secondary objectives are to compare maximal pain, consumption of supplementary analgesics, and the duratin of sensory block between groups.

DETAILED DESCRIPTION:
data will be collected on patient records and will be compared between groups of regional anesthesia.

Data will be :

* time to first analgesic request
* sensory block
* rescue analgesia during the first 24 hours after surgery
* maximal pain score during the first 24 hours after surgery
* patient satisfaction of managing care

ELIGIBILITY:
Inclusion Criteria:

- All adults patients scheduled for hand or wrist ambulatory surgery since 2016

Exclusion criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults patients scheduled for hand or wrist ambulatory surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
duration of analgesia | 24 hours
  time to first rescue analgesic request (opioid)

SECONDARY OUTCOMES:
maximal pain score during the first 24 hours after surgery | 24 hours
  Pain assessments during first 24 hours : maximal pain score during the first 24 hours after surgery
total rescue analgesia amounts the first 24 hours after surgery | 24 hours
  Pain assessments during first 24 hours : total rescue analgesia amounts the first 24 hours after surgery
duration of sensory block | 24 hours
  Pain assessments during first 24 hours : duration of sensory block

CONTACTS AND LOCATIONS:
Overall Officials: olivier CHOQUET, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC